CLINICAL TRIAL: NCT04193345
Title: The Maternal and Neonatal Impact of Early Versus Delayed Umbilical Cord Clamping Among Pregnant Severe Preeclampsia Patients Delivered by Cesarean Section
Brief Title: The Impact of Early Versus Delayed Umbilical Cord Clamping in Preeclamptic Pregnant Patients During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moutaz Sherbini, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MD-74-2019
Record Dates: First submitted 2019-12-08; First posted 2019-12-10 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Umbilical Cord Clamping
Keywords: Delayed Umbilical Cord Clamping; Preeclamptic Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early cord clamping (Active Comparator): The umbilical cord will be clamped within 15 seconds from delivery of the baby
  Interventions: Other: Documentation of Maternal blood loss and neonatal outcome
- Delayed cord clamping (Active Comparator): The umbilical cord will be clamped after 60 seconds from delivery of the baby
  Interventions: Other: Documentation of Maternal blood loss and neonatal outcome

INTERVENTIONS:
Other: Documentation of Maternal blood loss and neonatal outcome — Comparing and monitoring the maternal blood loss and neonatal effect of delayed umbilical cord clamping and early umbilical cord clamping after delivery of the baby durin cesarean delivery in severe preeclampsia

SUMMARY:
To compare the different maternal and neonatal impacts of early versus delayed umbilical cord clamping among pregnant preeclamptic patients delivered by cesarean section

DETAILED DESCRIPTION:
The study will include 62 pregnant women attending for severe preeclampsia and cesarean delivery will be done at the Kasr Elaini hospital (faculty of medicine - Cairo university).

Informed written consent: after discussing the nature of the study as well as the expected value, outcome, and possible adverse effects.

Full medical history: including full obstetric history and current pregnancy history (entailing the 1st day of LMP).

Thorough Clinical Examination: general (maternal body weight and vital signs) and full obstetric examination.

Obstetric ultrasonography: to confirm gestational age and the eligibility of the current pregnancy to participate in the study.

Preoperative laboratory tests: including prothrombin time, prothrombin concentration, complete blood count, and liver and kidney function tests.

Group allocation: On the day of the scheduled surgery, participants will be randomly and equally assigned into two groups; early clamping group n= 31 ( umbilical cord to be clamped within 15 s ) and delayed clamping group , n= 31 ( umbilical cord to be clamped at 60 sec ) , In all groups , Neonates will be held in a sterile towel or blanket below the level of the incision on maternal abdomen or between her legs at cesarean section. Care was taken that no tension or traction was placed on the cord. A stopwatch was used to mark the time , patients will receive an intravenous bolus of 5 IU oxytocin (Syntocinon, Novartis, Basel, Switzerland) and 20 IU oxytocin in 500 mL lactated Ringer's solution (infused at a rate of 125 mL/h) following the delivery of the baby All cesarean sections will be done under spinal anesthesia by an assistant lecturer and the following operative steps: pfannenstiel incision, transverse lower uterine segment incision, early cord clamping (< 15 seconds) or delayed cord clamping (after 60 sec) and the placenta will be removed by controlled cord traction after its spontaneous separation, closure of uterus in 2 layers, closure of anterior abdominal wall in anatomical manner (adequate hemostasis will be ensured in all operative steps).

The number and the difference of weight of operative towels (before and after LSCS) and amount of blood in suction unit will be recorded.

A complete blood count test will be performed 12 hours after delivery. neonatal laboratory results (hemoglobin and hematocrit, )will be collected within 4 hours of age, initial serum bilirubin was collected at 12 hours of age then to be repeated at day 3 for follow up.

Estimated Blood Loss (EBL) will be evaluated as follows:

A. The number of operative towels used. B. The difference of weight of operative towels (before and after cs) plus the amount of blood in suction unit (we will calculate 1 gram of weight difference equal to 1 ml blood loss).

C. EBL calculation according to the following formula:

EBL= EBV x Preoperative hematocrit- Postoperative hematocrit Postoperative hematocrit Where EBV is estimated blood volume of the patient in mL (equals weight in kg × 85).

The neonates clinical data, as APGAR Score, blood pressure, temperature, jaundice, pallor and cyanosis and respiratory distress syndrome will be collected by the attending neonatologist .All patients will be followed up following the delivery as regard occurrence of primary postpartum hemorrhage (within the first 24 hours), the need for blood transfusion (within the first 24 hours).

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women candidate for LSCS.
2. Age: 20-40 years old.
3. Maternal severe preeclampsia
4. CS under spinal anesthesia.
5. Singleton pregnancy

Exclusion Criteria:

1. Fetal death (IUFD).
2. Intrapartum surgical complications ( uterine artery injury or lower segment extension)
3. Medical disorders such as Diabetes mellitus or severe anemia
4. The need for immediate resuscitation like meconium aspiration .
5. Abnormal placentation or placental abruption
6. Liquor abnormalities ; oligo hydramnios
7. Anomalous fetus

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
the intra operative maternal blood loss | 24 hours
  To compare the early versus of delayed cord clamping on intra operative blood loss in pregnant patients diagnosed with severe preeclampsia

SECONDARY OUTCOMES:
the neonatal outcome | 4 days
  To compare the neonatal benefit from delayed cord clamping group versus early clamping in patients with severe preeclampsia during cesarean delivery
The incidence of post partum hemorrhage | 24 hours
  To assess the extra need for ecbolics and the actual incidence of post partum hge with both methods

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rashwan A, Eldaly A, El-Harty A, Elsherbini M, Abdel-Rasheed M, Eid MM. Delayed versus early umbilical cord clamping for near-term infants born to preeclamptic mothers; a randomized controlled trial. BMC Pregnancy Childbirth. 2022 Jun 25;22(1):515. doi: 10.1186/s12884-022-04831-8. PMID 35752762
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/18425897
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/28002310
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/24150027
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/22895933